CLINICAL TRIAL: NCT05545943
Title: Effects of 2-day and 6-day Calorie Restriction and Whole-body Cooling Strategies on Health-related Indicators, Cognitive and Motor Functions
Brief Title: Effects of Calorie Restriction and Cold Stimuli on Health-related Indicators, Cognitive and Motor Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: LithuanianSportsU-10
Record Dates: First submitted 2022-09-09; First posted 2022-09-19 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Calorie Deficiency; Fasting; Cold Exposure
Keywords: cognition; motor function; metabolism; young adults; fasting; starvation; men; women; calorie deprivation; stress; kynurines; catecholamines; glucose tolerance; energy expenditure; weight loss
MeSH Terms: conditions — Fasting; Starvation; Multiple Endocrine Neoplasia Type 1; Weight Loss

STUDY DESIGN:
Intervention Model Description: This project consisted of two parts. For the first part was used randomized parallel model, and we aimed to investigate fasting duration effect, whereas for the second part was used randomized crossover model and we aimed to investigate if cold exposure can modify fasting evoked effects on health-related indicators, cognition and motor function.
Who Masked: Investigator
Masking Description: The researchers who analyzed the saliva and venous blood samples were blinded to the experimental conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 2-days of calorie restriction with whole body cooling (Experimental): Healthy young subjects participated in a 2-day CR (0 kcal with water provided ad libitum ) with two 10-min whole body cooling practices on separate days.
  All participants were asked to not perform excessive sports activities while the research was ongoing, not to be involved in any temperature-manipulation program or extreme temperature exposure for ⩾3 months; do not use any medications that could affect experimental data.
  Interventions: Other: 2-days of zero calorie restriction and whole-body cold-water immersion
- 6-days of calorie restriction (Experimental): Healthy young subjects participated in 6-day CR (0 kcal with water provided ad libitum).
  All participants were asked to not perform excessive sports activities while the research was ongoing, not to be involved in any temperature-manipulation program or extreme temperature exposure for ⩾3 months; do not use any medications that could affect experimental data.
  Interventions: Other: 6-days of calorie restriction
- 2-days of the usual diet (control) (No Intervention): During the control trial, the healthy young subjects were instructed to maintain their previous eating habits for 2 days.
  All participants were asked to not perform excessive sports activities while the research was ongoing, not to be involved in any temperature-manipulation program or extreme temperature exposure for ⩾3 months, CR programmes; do not use any medications that could affect experimental data.
- 6 days of the usual diet (control) (No Intervention): During the control trial, the healthy young subjects were instructed to maintain their previous eating habits for 6 days.
  All participants were asked to not perform excessive sports activities while the research was ongoing, not to be involved in any temperature-manipulation program or extreme temperature exposure for ⩾3 months, CR programmes; do not use any medications that could affect experimental data.
- 2-days of calorie restriction without whole-body cooling (Experimental): Healthy young subjects participated in a 2-day CR (0 kcal with water provided ad libitum ) without whole body cooling.
  All participants were asked to not perform excessive sports activities while the research was ongoing, not to be involved in any temperature-manipulation program or extreme temperature exposure for ⩾3 months; do not use any medications that could affect experimental data.
  Interventions: Other: 2-days of zero calorie restriction without whole-body cold-water immersion
- 2-days of usual diet with whole-body cooling (Active Comparator): Healthy young subjects participated two 10-min whole body cooling practices on separate days and were instructed to maintain their previous eating habits for 6 days.
  All participants were asked to not perform excessive sports activities while the research was ongoing, not to be involved in any temperature-manipulation program or extreme temperature exposure for ⩾3 months, CR programmes; do not use any medications that could affect experimental data.
  Interventions: Other: 2-days of usual diet with whole-body cold-water immersion

INTERVENTIONS:
Other: 2-days of zero calorie restriction and whole-body cold-water immersion — The 2-days (48 hours) of zero-calorie restricted diet (with water provided ad libitum) with two whole-body cold-water immersion sessions on separate days. During cooling procedures, the participant was immersed in 14° water bath in semi recumbent position up to the level of the manubrium for 10 min.
  Arms: 2-days of calorie restriction with whole body cooling
Other: 6-days of calorie restriction — The 6-days (144 hours) of prescribed zero-calorie prescribed diet with water provided ad libitum.
  Arms: 6-days of calorie restriction
Other: 2-days of zero calorie restriction without whole-body cold-water immersion — 2 days (48 hours) of prescribed zero-calorie diet with water provided ad libitum .
  Arms: 2-days of calorie restriction without whole-body cooling
Other: 2-days of usual diet with whole-body cold-water immersion — Two whole-body cold-water immersion sessions on separate days. During cooling procedures, the participant was immersed in 14° water bath in semi recumbent position up to the level of the manubrium for 10 min. During intervention, participants were instructed to maintain their previous eating habits.
  Arms: 2-days of usual diet with whole-body cooling

SUMMARY:
The goal of this clinical trial was to identify if duration of acute calorie restriction (CR)/fasting or combination CR with cold stimuli have any effects on mental and physical health-related markers, and to clarify if different fasting strategies have any effect on cognitive and motor functioning efficiency in different genders.

The main questions it aims to answer were:

* Does fasting duration have any effect on fasting evoked responses?
* Does cold interventions can modulate fasting evoked responses?
* Does sex have any effect on acute fasting evoked responses?

For the first part, participants were randomly classified into 4 groups: two experimental groups: 2-days of CR (0 kcal diet) and 6-days of CR (0 kcal diet), and two control groups: 2-days or 6-days usual diet. For the second part, participants were randomly assigned to undergo the following conditions: 2-days of CR with two 10-min whole-body cold-water immersions on separate days, 2-days of CR without cold-water immersion, 2-days without CR with two 10-min whole-body cold-water immersions on separate days, or 2-days of the usual diet without cold-water immersion in a randomized crossover fashion. Changes in anthropometric characteristics, perceived stress, metabolism, overall health (total blood count, sex hormones, etc.), psycho-emotional state, cognitive and motor functions were examined.

DETAILED DESCRIPTION:
The goal of this clinical trial was to identify if duration of acute calorie restriction (CR)/fasting or combination CR with cold stimuli have any effects on mental and physical health-related markers, and to clarify if different fasting strategies have any effect on cognitive and motor functioning efficiency in different genders.

At first study part, participants were randomly classified into 4 groups: two experimental groups: 2-days of calorie restriction (CR) (0 kcal diet) and 6-days of CR (0 kcal diet), and two control groups: 2-days or 6-days usual diet. In the experimental groups, the participants were instructed to follow a prescribed zero-calorie diet with water provided ad libitum over a period of 2 or 6 days. In the control groups, the participants were instructed to maintain their previous eating habits for 2 or 6 days. Body weight and composition, heart rate variability, pulmonary gas exchange, blood pressure, and body temperature were assessed. Subsequently, participants completed self-assessment questionnaires, and then saliva samples were collected for further cortisol and sex hormones analysis, also capillary and venous blood samples were taken for ketone, glucose, insulin, lipid profile, catecholamines, brain-derived neurotrophic factor, total antioxidant capacity, malondialdehyde, glucagon, interleukin-10, metabolites of the kynurenines pathway and complete blood count concentrations evaluation. Then, the manual dexterity, and the cognitive and neuromuscular functions were assessed. The same measurements were repeated before each trial, after each trial and after 1 week.

At second part, participants were randomly assigned to undergo the following conditions: 2-days of CR with two 10-min whole-body cold-water immersions on separate days, 2-days of CR without cold-water immersion, 2-days without CR with two 10-min whole-body cold-water immersions on separate days, or 2-days of the usual diet without cold-water immersion in a randomized crossover fashion. The same measurements described in first part were repeated before each and after each condition.

ELIGIBILITY:
Inclusion criteria:

* body mass index 19.5-29.9 kg/m2,
* age 18-40 years,
* no excessive regular moderate or vigorous physical activity, i.e., ≥3 times per week,
* non-smokers,
* no medications that could affect the results of experiment,
* no history of any eating, oncological, metabolic, cardiovascular, skeletal, neuromuscular, pulmonary disorders or diseases, mental disabilities or conditions that could be worsened by exposure to acute cold (14°) water or fasting and affect experimental variables,
* no history of alcoholism or dependence on psychotropic drugs,
* no blood/needle phobia,
* no involvement in any temperature-manipulation program or extreme temperature exposure for ⩾3 months,

Exclusion criteria: smoking, were in a weight-reduction program, followed a low-carbohydrate diet.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Change in body mass and body composition (kg) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Body mass and composition (in kg) was evaluated using Tanita Body Composition Analyzer (Japan).
Change in body mass index (kg/m2) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  The body mass index (in kg/m2) was defined as the body mass divided by the square of the body height.
Change in substrate oxidation | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Oxygen consumption and carbon dioxide output every 5 s on a breath-by breath basis using an Oxycon Mobile spirometry system (Oxygen Mobile, Jaeger/ VIASYS Healthcare, Germany) was measured at rest, and the respiratory quotient (RQ=VCO2/VO2) was computed to determine substrate utilisation. The RQ values for fat was assumed as 0.7, for protein was assumed as 0.8 and for carbohydrate was assumed as 1.0.
Change in energy expenditure (kcal/day) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Resting energy expenditure (REE) using Weir equation modified Weir equation: REE (kcal/day)=[3.941(oxygen consumption) + 1.106(carbon dioxide output)] x 1440
Change in body temperature (°C) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Rectal temperature (°C) was measured using a thermocouple (Rectal Probe, Ellab, Denmark) inserted to a depth of 12 cm past the anal sphincter, skin temperature (°C) was measured with thermistors (Skin/Surface Probe, DM852, Ellab) at three sites: back, thigh, and forearm, and right lateral gastrocnemius muscle temperature (°C) was measured using a needle microprobe (MKA; Ellab).
Change in heart rate variability (ms) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  R-R intervals (in ms) in supine resting conditions were recorded using a Polar HR sensor (Finland) and and simultaneously transferred to Polar Pro Trainer 5 software (Finland).
Change in heart rate variability (time domain) (ms) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Heart rate variability data were analyzed using Kubios HR Variability Analysis software (Finland). In the time domain that reflects general heart rate variability (HRV), the standard deviation of normal-to-normal intervals (SDNN; estimate of overall HRV) and the root mean square of successive differences (RMSSD; estimate of short-term components of HRV) were assessed (in ms).
Change in heart rate variability (time domain) (Ln) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Heart rate variability data were analyzed using Kubios HR Variability Analysis software (Finland). In the time domain that reflects general heart rate variability (HRV), the standard deviation of normal-to-normal intervals (SDNN; estimate of overall HRV) and the root mean square of successive differences (RMSSD; estimate of short-term components of HRV) were assessed and logarithmically transformed (Ln) to correct the skewness of distribution.
Change in heart rate variability (frequency domain) (ms2) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Heart rate variability data were analyzed using Kubios HR Variability Analysis software (Finland). In the frequency domain that measures the more specific contribution of the autonomic nervous system branch, we used the fast Fourier transform to assess low-frequency (LF; estimates sympathetic and parasympathetic activity) and high-frequency (HF; estimates parasympathetic activity) powers in absolute units (in ms2).
Change in heart rate variability (frequency domain) (Ln) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Heart rate variability data were analyzed using Kubios HR Variability Analysis software (Finland). In the frequency domain that measures the more specific contribution of the autonomic nervous system branch, we used the fast Fourier transform to assess low-frequency (LF; estimates sympathetic and parasympathetic activity) and high-frequency (HF; estimates parasympathetic activity) powers were assessed and logarithmically transformed (Ln) to correct the skewness of distribution.
Change in heart rate variability (frequency domain) (nu) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Heart rate variability data were analyzed using Kubios HR Variability Analysis software (Finland). In the frequency domain that measures the more specific contribution of the autonomic nervous system branch, we used the fast Fourier transform to assess low-frequency (LF; estimates sympathetic and parasympathetic activity) and high-frequency (HF; estimates parasympathetic activity) powers in normalized units (in nu).
Change in heart rate (bpm) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Heart rate (in bpm) was recorded using a heart rate sensor with a chest strap (Polar, Finland) in laying position at rest.
Change in blood pressure (mmHg) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Resting systolic and diastolic blood pressure (in mmHg) was measured using a digital electronic blood pressure monitor (Microlife, Switzerland)
Change in perceived stress | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Perceived stress was evaluated with visual analog scales (VAS) ranging from 0 ("no stress") to 100 ("the highest stress imaginable").according to how participants feel "right now".
Change in appetite sensations | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Appetite sensations (hunger and fullness) were evaluated with VAS ranging from 0 ("I am not hungry at all/not at all full") to 100 ("I have never been more hungry/totally full") according to how participants feel "right now".
Change in mood state | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Mood state was evaluated with Brunel mood scale according to how participants feel "right now". The scale consists of 24 items divided into six subscales: anger, confusion, depression, fatigue, tension, and vigor. The items are answered on a 5-point scale, and each subscale, with four relevant items, are summed to produce a raw score in the range of 0-16, where a higher score indicates greater endorsement of the specific mood state.
Change in venous complete blood count (10^9/L) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Venous complete blood count with 5 different white blood count (WBC) components (absolute neutrophils, lymphocytes, monocytes, eosinophils, basophils) analysis (in 10^9/L) was performed using an automated Mythic 60 hematology analyzer (Switzerland).
Change in venous complete blood count (%) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Venous complete blood count with 5 different white blood count (WBC) components (absolute neutrophils, lymphocytes, monocytes, eosinophils, basophils) analysis (in %) was performed using an automated Mythic 60 hematology analyzer (Switzerland).
Change in serum female sex hormones concentration (pg/mL) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  The venous serum 17beta-estradiol and progesterone (in pg/mL) were measured using enzyme-linked immunosorbent assay kits and a Spark multimode microplate reader (Tecan, Austria).
Change in serum female sex hormones concentration (mIU/ml) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  The venous serum follicle stimulating and luteinizing hormones (in mIU/ml) were measured using enzyme-linked immunosorbent assay kits and a Spark multimode microplate reader (Tecan, Austria).
Change in serum brain-derived neurotrophic factor concentration (pg/ml) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  The venous serum brain-derived neurotrophic factor (in pg/ml) was measured using enzyme-linked immunosorbent assay kits (Cat.No. DBD00; R&D Systems, Emeryville, USA) and a Spark multimode microplate reader (Tecan, Austria).
Change in serum interleukin-10 concentration (pg/ml) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  The venous serum interleukin (in pg/ml) was measured using enzyme-linked immunosorbent assay kits (Cat. No. 30147233; IBL International GmBH, Germany) and a Spark multimode microplate reader (Tecan, Austria).
Change in serum insulin concentration (μIU/ml) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  The venous serum insulin concentrations (in μIU/ml) were measured using enzyme-linked immunosorbent assay kits (Cat. No. E-EL-H2237, Elabscience, China) and a Spark multimode microplate reader (Tecan, Austria).
Change in serum glucagon concentration (pg/ml) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  The venous serum glucagon concentrations (in pg/ml) were measured using enzyme-linked immunosorbent assay kits (DIAsource ImmunoAssays S.A.,Belgium) and a Spark multimode microplate reader (Tecan, Austria).
Change in plasma catecholamines concentration (ng/ml) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  The venous plasma adrenaline and noradrenaline concentrations (in ng/ml) were measured using enzyme-linked immunosorbent assay kits (Cat. No. RE59242, IBL International GmbH, Germany) and a Spark multimode microplate reader (Tecan, Austria).
Change in plasma malondialdehyde concentration (nmol/ml) | Pre-condition, 48, 84 and 144 hours post-condition, and 1 week after recovery
  The venous plasma malondialdehyde concentrations (in nmol/l) were measured using a solid phase nzyme-linked immunosorbent assay (Cat. No. E1371Hu, Bioassay Technology Laboratory, Shangai, China) and a Spark multimode microplate reader (Tecan, Austria).
Change in plasma total antioxidant capacity (mmol/l) | Pre-condition, 48, 84 and 144 hours post-condition, and 1 week after recovery
  The venous plasma total antioxidant capacitys (in mmol/l) were measured colorimetrically with an assay kit (Cat. No.E-BC-K271-M, Elabscience Biotechnology Inc, Houston, USA) and using a Spark multimode microplate reader (Tecan, Austria).
Change in venous glucose concentration (mmol/l) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  The venous glucose concentration (in mmol/l) was measured in venous blood samples using a Glucocard X-mini plus glucose analyser (Arkray, Japan).
Change in insulin sensitivity | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  An oral glucose insulin sensitivity [OGIS] index derived from an oral glucose tolerance test was calculated.
Change in plasma metabolites of the kynurenine pathway (μm) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  An ultra-performance liquid chromatography-tandem mass spectrometry system (UPLC-MS/MS) to measure venous plasma levels of tryptophan, kynurenine, kynurenic acid, 3-hydroxy-kynurenine, quinolinic acid, nicotinamide and picolinic acid (in μm). The UPLC-MS/MS system used a Xevo TQ-XS triple quadrupole mass spectrometer (Waters) with a Z-spray electrospray interface, and the system was operated in electrospray positive multiple reaction monitoring mode.
Change in salivary cortisol concentration (µg/dl) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  The saliva samples were collected to measure cortisol level (in µg/dl) using a enzyme-linked immunosorbent assay (ELISA) kits and a Spark multimode microplate reader (Tecan, Austria).
Change in salivary testosterone concentration (µg/dl) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  The saliva samples were collected to measure testosterone level (in µg/dl) using a enzyme-linked immunosorbent assay (ELISA) kits and a Spark multimode microplate reader (Tecan, Austria).
Change in capillary lipid profile (mmol/l) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  The capillary blood samples were collected from finger to measure lipid profile (in mmol/l) (total cholesterol, high density and low density cholesterol, triglycerides) using a CardioChek PA analyzer (USA).
Change in manual dexterity performance (sec) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  The Grooved Pegboard was used to evaluate the ability to coordinate the fingers and manipulate objects promptly in time twice (in sec).
Change in information processing (μV) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Using a 32-channel Standard Brain Cap (EasyCap GmbH, Germany), event-related potentials (ERPs) during oddball tasks by two modalities (auditory and visual) were recorded. Peak amplitudes (μV) of the N1, N2 and P3 at three sites (Fz, Cz, and Pz) were defined.
Change in information processing (ms) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Using a 32-channel Standard Brain Cap (EasyCap GmbH, Germany), event-related potentials (ERPs) during oddball tasks by two modalities (auditory and visual) were recorded. Latencies (ms) of the N1, N2 and P3 at three sites (Fz, Cz, and Pz) were defined.
Change in brain neural network activity (µV2) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Resting electroencephalography was recorded using a 32-channel Standard Brain Cap (EasyCap GmbH, Germany). Participant's data were averaged across the epochs for Fz, Cz and Pz electrodes, and mean absolute power (in µV2) was computed for theta (4-8 Hz), alpha (8-12 Hz) and beta (12-30 Hz) frequency band.
Change in cognitive performance (ms) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Two oddball tasks were used in this study: in one task, visual stimuli were presented, and in the other task, auditory stimuli were presented. Reaction times (in ms) were measured.
Change in cognitive performance (%) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Two oddball tasks were used in this study: in one task, visual stimuli were presented, and in the other task, auditory stimuli were presented. Accuracy of response to the target stimulus (in %) were measured.
Change in reflexes (mV) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Soleus H-reflexes, V-waves and M-waves were evoked by 0.5 ms square-wave pulses using a high-voltage stimulator (Digitimer, UK). The amplitudes (in mV) of the electrical evoked reflexes were evaluated.
Change in reflexes (ms) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Soleus H-reflexes, V-waves and M-waves were evoked by 0.5 ms square-wave pulses using a high-voltage stimulator (Digitimer, UK). The latencies (in ms) of the electrical evoked reflexes were evaluated.
Change in muscle activity (mV) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Tibial muscles electromyographic (EMG) amplitude (in mV) parameters of muscular activity were measured using surface EMG (Biometrics, UK) thorough neuromuscular function assessment.
Change in muscle activity (Hz) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Tibial muscles electromyographic (EMG) frequency (in Hz) parameters of muscular activity were measured using surface EMG (Biometrics, UK) thorough neuromuscular function assessment.
Change in voluntary torque (Nm) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Isometric and isokinetic voluntary torques (in Nm) of the ankle plantar flexion/dorsiflexion muscles were measured using an isokinetic dynamometer (Biodex Medical Systems, USA).
Change in involuntary torque (Nm) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Involuntary torque of the ankle plantar flexion muscles were measured using an isokinetic dynamometer (Biodex Medical Systems, USA) and a high-voltage stimulator (Digitimer DS7A, Digitimer, UK). Peak torques (in Nm) induced by electrical stimulation at 20 Hz,at 100 Hz, and at TT100 were measured.
Change in muscle contraction and relaxation (ms) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  The contraction and half-relaxation time (in ms) were measured in resting TT100 contractions.
Change in central activation ratio (%) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  To evaluate central activation ratio (CAR), a TT-100 Hz stimuli was superimposed on the maximal voluntary contraction (MVC), and the CAR was computed using the following equation: CAR = MVC/(MVC+TT-100 Hz) × 100%, where where a CAR of 100% indicates complete activation of the exercising muscle and a CAR < 100% indicates central activation failure or inhibition.
Change in reactive strength | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  The drop jump test on a force mobile platform (AccuPower, AMTI, USA) was used to evaluate reactive-strength. Jumps were performed while holding the hands of the subject on the hips were requested jump as fast as possible after the drop off from the platform and make sure that the jump is the highest possible. Reactive strength index as jump height / time to take off was calculated.
Change in jump performance (cm) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  The drop jump test on a force mobile platform (AccuPower, AMTI, USA) was used to evaluate jump performance. Jumps were performed while holding the hands of the subject on the hips were requested jump as fast as possible after the drop off from the platform and make sure that the jump is the highest possible. Jump height (in cm) height was evaluated.
Change in jump performance (m/s) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  The drop jump test on a force mobile platform (AccuPower, AMTI, USA) was used to evaluate jump performance. Jumps were performed while holding the hands of the subject on the hips were requested jump as fast as possible after the drop off from the platform and make sure that the jump is the highest possible. Time to take off (in m/s) was evaluated.

SECONDARY OUTCOMES:
Change in height (m) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Height (in m) was measured using a Harpenden anthropometer set (Holtain Ltd, UK)
Change in skinfold thickness (mm) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Skinfolds thickness (in mm) was measured using a skinfold caliper (Saehan, Korea) at 7 sites: chest, midaxilla, triceps, subscapular, abdominal, suprailiac and thigh.
Change in body fatness (%) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  7-Site Skinfold Jackson & Pollock protocol was used to estimate body fat (in %) based on measurements of subcutaneous fat. As presented earlier, skinfolds were measured at 7 sites, and further body fatness was calculated as 495/(1.112-(0.00043499*s(sum of 7 skinfolds)+(0.00000055*s*s)-(0.00028826*a(age)))-450 for males and 495/(1.097-(0.00046971*s)+(0.00000056*s*s)-(0.00012828*a))-450 for females.
Change in physical activity (Step count) | 3 days before condition, during 48 or 144 hours of interventions and during 1 week post-condition. (2 weeks)
  Garmin activity tracker estimated the step count.
Change in sleep (h) | 3 days before condition, during 48 or 144 hours of interventions and during 1 week post-condition. (2 weeks)]
  Sleep statistics including total hours of sleep and the time spent in different sleep stages were assessed with Garmin activity tracker.
Change in oxygen consumption and carbon dioxide output (ml/min) | Pre-condition, 48 or 144 hours post-condition, and 1 week after recovery
  Oxygen consumption and carbon dioxide output (in ml/min) every 5 s on a breath-by breath basis using an Oxycon Mobile spirometry system (Oxygen Mobile, Jaeger/ VIASYS Healthcare, Germany) was measured at rest.
Change in capillary blood ketone concentrations (mmol/l) | Pre-condition, 24, 48 or 144 hours post-condition, and 1 week after recovery
  The capillary blood ketone concentration (in mmol/l) was assessed using an Abbott FreeStyle Optium Neo H blood glucose and ketone monitoring system (Australia) using blood obtained from a finger-prick sample.
Change in capillary blood glucose concentrations (mmol/L) | Pre-condition, 24, 48 or 144 hours post-condition, and 1 week after recovery
  The capillary blood glucose concentration (in mmol/L) was assessed using an Abbott FreeStyle Optium Neo H blood glucose and ketone monitoring system (Australia) using blood obtained from a finger-prick sample.

CONTACTS AND LOCATIONS:
Overall Officials: Katerina Židonienė, Principal Investigator — Lithuanian Sports University
Locations (1):
- Lithuanian Sports University, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Solianik R, Zidoniene K, Baranauskiene N, Brazaitis M. Fasting for 48 h induced similar glucose intolerance in both sexes despite greater perceived stress and decreased estradiol levels in females. Eur J Appl Physiol. 2024 May;124(5):1449-1459. doi: 10.1007/s00421-023-05378-y. Epub 2023 Dec 18. PMID 38108909